CLINICAL TRIAL: NCT06480630
Title: Effectiveness and Safety of a Single-Center Clinical Study on a CD25 Monoclonal Antibody-Containing GVHD Prophylaxis Scheme to Reduce the Incidence of Severe Acute GVHD After Umbilical Cord Blood Transplantation for Malignant Hematologic Diseases
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Anhui Provincial Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CD25-2024
Record Dates: First submitted 2024-06-25; First posted 2024-06-28 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Acute Graft Versus Host Disease; Malignant Hematologic Neoplasm
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Basiliximab

STUDY DESIGN:
Intervention Model Description: Addition of CD25 monoclonal antibody at +3 days post unrelated umbilical cord blood transplantation (UCBT)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- basiliximab group (Experimental)
  Interventions: Drug: Basiliximab

INTERVENTIONS:
Drug: Basiliximab — Addition of CD25 monoclonal antibody（Basiliximab） at +3 days post unrelated umbilical cord blood transplantation (UCBT)

SUMMARY:
Evaluating the safety and effectiveness of a CD25 monoclonal antibody-based prophylactic acute graft-versus-host-disease (aGVHD) regimen following unrelated umbilical cord blood transplantation (UCBT) for malignant hematologic disorders in reducing severe aGVHD.

DETAILED DESCRIPTION:
Acute graft-versus-host disease (aGVHD) is a major complication and leading cause of non-relapse mortality following allogeneic hematopoietic stem cell transplantation (allo-HSCT). Preliminary research findings suggest that the addition of CD25 monoclonal antibody at +3 days post unrelated umbilical cord blood transplantation (UCBT) has reduced the incidence of grade III-IV aGVHD compared to previous protocols. In order to further explore how to improve prevention strategies of aGVHD and reduce the incidence of severe aGVHD, we performed this study to evaluate the safety and effectiveness of a prophylactic GVHD regimen utilizing CD25 monoclonal antibody post-UCBT for malignant hematologic disorders, aimed at reducing the incidence of severe aGVHD.

ELIGIBILITY:
Inclusion Criteria:

* Malignant hematologic disorders;
* Patients undergoing UCBT;
* Female patients of childbearing potential must have a negative pregnancy test and agree to use effective contraception during treatment and for the following year.

Exclusion Criteria:

* Non-malignant hematologic disorders;
* History of allogeneic hematopoietic stem cell transplantation or solid organ transplantation;
* Uncontrolled bacterial, viral, or fungal infections. "Uncontrolled" is defined as lack of clinical improvement or progression despite adequate antimicrobial therapy;
* HIV infection or active hepatitis B or C virus infection;
* Pregnant or lactating women;
* Substance abusers; subjects with uncontrolled psychiatric disorders; individuals with cognitive dysfunction;
* Participation in similar clinical studies within the past 3 months;
* Subjects deemed unsuitable by the investigator (e.g., those expected to be unable to adhere to treatment due to financial constraints).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
The cumulative incidence of grade III-IV acute graft-versus-host disease (aGVHD) | within 100 days post-UCBT
  The primary endpoint of the study will be the development of aGVHD in the first 100 days post-transplant. Acute GVHD was graded according to the International Consortium criteria.

SECONDARY OUTCOMES:
The incidence rate and occurrence time of pre-engraftment syndrome (PES) | within 30 days post-UCBT
  The occurrence time and cumulative incidence of PES within 30 days post-UCBT. The PES was diagnosed according to the criteria of engraftment syndrome (ES) .
The cumulative incidence of neutrophil engraftment at 28 days after transplantation | within 28 days post-UCBT
  Neutrophil engraftment time was defined as the first of three consecutive days during which the neutrophil count was at least 0.5×10^9/L.
The cumulative incidence of platelet engraftment at 100 days after transplantation | within 100 days post-UCBT
  Platelet engraftment is defined as independence from platelet transfusion for at least 7 days with a platelet count of more than ≥ 20 × 10^9/L.
The incidence of grade II to IV aGVHD | within 100 days post-UCBT
  The cumulative incidence of grade II to IV aGVHD in the first 100 days post-transplant. aGVHD was graded according to the aGVHD International Consortium criteria.
The cumulative incidence of chronic GVHD at 360 days after transplantation | 360 days
  The severity of chronic GVHD was graded according to the 2014 NIH criteria.
The cumulative incidence of transplant-related mortality at 180 days after transplantation | 180 days
  The cumulative incidence of transplant-related mortality at 180 days after transplantation.
The cumulative incidence of relapse | 1 year
  The cumulative incidence of relapse at 1 year after transplantation.
The probability of disease-free survival(DFS) | 1 year
  The DFS was defined as the interval between transplantation and disease recurrence, death or the last follow-up date, whichever occurred first.
The probability of overall survival(OS) | 1 year
  The OS was determined to be the time from the first day of transplantation until death from any cause or the last follow-up date.
The probability of GVHD-free, relapse-free survival(GRFS) | 1 year
  The composite endpoint of GRFS was defined as the first events occurring after transplantation among Grade III to IV aGVHD, moderate to severe cGVHD, relapse, or death for any reason.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoyu Zhu, Ph.D, Principal Investigator — The First Affiliated Hospital of USTC (Anhui Provincial Hospital)
Locations (1):
- The First Affiliated Hospital of University of Science and Technology of China (Anhui Provincial Hospital), Hefei, China

IPD SHARING:
Plan to Share IPD: No